CLINICAL TRIAL: NCT03739047
Title: The Impact of Desensitization as a Modality to Reduce Oral Hypersensitivity and Improve Intake in Children With Pediatric Feeding Disorders
Brief Title: Desensitization to Reduce Oral Hypersensitivity and Improve Intake for Children With Feeding Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Natalie Morris, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00143299
Record Dates: First submitted 2018-10-29; First posted 2018-11-13 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Feeding Disorder
Keywords: Children with feeding disorders
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Desensitization, Psychologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desensitization with flipped spoon (Experimental): Children in this study will receive behavioral feeding treatment. This arm will include desensitization.
  Interventions: Behavioral: Desensitization with flipped spoon
- flipped spoon (Placebo Comparator): Children in this study will receive behavioral feeding treatment.
  Interventions: Behavioral: flipped spoon

INTERVENTIONS:
Behavioral: Desensitization with flipped spoon — Both groups will begin with a baseline phase: escape extinction (non-removal of an upright small maroon spoon) plus continuous access to reinforcement. The baseline phase will take place for 3, 5-bite sessions or until the data become stable. The baseline phase will be followed by desensitization. Desensitization will be conducted for 3, 45-minute treatment meals. Puree will be presented on a flipped EZ spoon after the desensitization sessions are completed. Bite size will be gradually increased. Acceptance of an upright EZ spoon and eventually an upright maroon spoon will be probed based on stability of the data.
  Arms: Desensitization with flipped spoon
Behavioral: flipped spoon — Both groups will begin with a baseline phase: escape extinction (non-removal of an upright small maroon spoon) plus continuous access to reinforcement. The baseline phase will take place for 3, 5-bite sessions or until the data become stable. The baseline phase will be followed by puree being presented from a flipped EZ spoon. Bite size will be gradually increased. Acceptance of an upright EZ spoon and eventually an upright maroon spoon will be probed based on stability of the data.
  Arms: flipped spoon

SUMMARY:
Many children with feeding disorders frequently gag, vomit, spit out their food, and/or hold food in their cheeks. These behaviors make it difficult for children to eat enough food to grow. The purpose of this study is to evaluate if a specific behavioral feeding intervention called desensitization is an effective intervention to improve oral intake in children with feeding disorders by decreasing gagging, vomiting, spitting, and holding food in the cheeks. The study will enroll eligible children (6) and their caretakers (6) in the study and they will receive behavioral feeding treatment. All treatment sessions will be videotaped and the study will last a maximum 8 weeks after the first treatment visit, or until treatment goals have been met.

DETAILED DESCRIPTION:
Children with complex medical histories may have limited, delayed, or no early oral feeding experiences, which decreases the likelihood of independently developing appropriate oral motor skills required for eating. Children who are introduced to solid foods after 6-7 months of age frequently gag, choke, or vomit due to inefficient oral-motor skills. In typically developing children, gagging weakens as a child learns to chew around 7-months of age. However, children with feeding disorders do not have the same opportunities to weaken the natural gag reflex due to limited experience with oral feedings. As a result, they often become hypersensitive to any tactile stimulation and averse to foods and utensils touching specific parts of the mouth. There is a gap in the behavioral feeding literature addressing oral hypersensitivity and behaviors that interfere with swallowing (i.e., packing, expelling, gagging, vomiting). Some work surrounding desensitization of the oral cavity has already been done within other disciplines (i.e., occupational therapists and speech and language pathologists); however, desensitization has not been well-defined, nor has it been empirically studied.

(1) Specific Aims: The proposed study is designed to assess the following aims:

1. Define an oral-desensitization protocol to improve oral intake and decrease gags and emesis in children with feeding disorders.
2. Evaluate the efficacy of the brief implementation of an oral-desensitization protocol alone and in combination with the antecedent-based procedure, flipped spoon.
3. To explore the relationship between behavioral feeding intervention and child oral and motor proficiency.
4. To explore the relationship between behavioral feeding intervention and parent and child outcomes including parenting stress, mealtime feeding behaviors, and general child behavioral functioning.

(2) Research Hypotheses: The proposed study is designed to test the following hypotheses:

* Effect of flipped spoon versus flipped spoon + desensitization. It is hypothesized that there will be a faster decrease in (1) gags, (2) latency to clean mouth, (3) packs, (4) emesis, and (5) CI's with those participants who receive oral desensitization prior to the flipped spoon intervention. It is also hypothesized that children who receive desensitization prior to flipped spoon will be able to transition back to an upright spoon more quickly when compared to children who did not receive desensitization.
* Effect of behavioral feeding intervention on child oral and motor proficiency. Exploratory analyses will be conducted to examine pre-test and post-test ratings of child oral and motor proficiency. It is anticipated that the oral-motor coordination of the participants will significantly improve.
* The relationship between behavioral feeding intervention and parent/child outcomes. Exploratory analyses will be conducted to examine pre-test and post-test ratings of parenting stress, mealtime feeding behaviors, and general child behavioral and emotional functioning. It is anticipated that parent-reported ratings in these areas will improve from pre-test to post-test.

Treatment:

Participants will be randomly assigned to one of two treatment groups: desensitization + traditional behavioral intervention or traditional behavioral intervention alone. All participants will be treated for a maximum of 40 treatment days, or until treatment goals have been met. A total of 3, 45-minute meals will be held each day for a total of 120 meals throughout treatment. Trained feeding therapists from the Interdisciplinary Pediatric Feeding Program at Mott Children's Hospital will conduct sessions in treatment rooms with one-way mirrors. Caregivers will be given the option to observe through the one-way mirror or stay in the treatment room with the participant. The behavioral intervention will involve a combination of escape extinction and antecedent manipulation of the food (e.g., limiting bite size, using a flipped spoon to deposit the bolus). The behavioral intervention plus desensitization will include the above in addition to desensitization of the oral cavity. Desensitization will occur for the first 3 meals. This involves systematically stimulating different areas of the oral cavity (cheeks, palate, tongue, sides of tongue) to provoke and ultimately decrease the gag response allowing eating to be easier for participants. Data will be collected throughout each meal. All feeding sessions will be recorded to ensure protocol fidelity and for the purposes of collecting reliability data.

ELIGIBILITY:
Inclusion Criteria:

* Behavior problems (i.e., spitting, crying, head turning, gagging, physical aggression) are interfering with feeding
* Medical causes of feeding disorder have been treated or are well-controlled without resolution of the feeding problem
* Normal feeding milestones have not been met or regression has occurred
* Enteral feeding dependence as defined by the participant relying on Nasal Gastric or gastrostomy-tube feedings in order to receive appropriate nutrition and gain weight
* Accepts a limited number of foods and limited volume of foods by mouth (i.e., not enough variety or volume to maintain growth and/or good nutritional status)

Exclusion Criteria:

* Children who had anatomical/active medical problems that prohibit safe oral intake will be excluded

Ages: 10 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline frequency of gags at 8 weeks, or when treatment goals are met | Baseline, up to eight weeks after first treatment visit
  Participants will be observed for gags to evaluate the effectiveness of Desensitization
Change from baseline latency to clean mouth at 8 weeks, or when treatment goals are met | Baseline, up to eight weeks after first treatment visit
  Participants will be observed for latency to clean mouth to evaluate the effectiveness of Desensitization
Change from baseline frequency of packs at 8 weeks,or when treatment goals are met | Baseline, up to eight weeks after first treatment visit
  Participants will be observed for number of packs to evaluate the effectiveness of Desensitization
Change from baseline frequency of emesis at 8 weeks, or when treatment goals are met | Baseline, up to eight weeks after first treatment visit
  Participants will be observed for emesis to evaluate the effectiveness of Desensitization
Change from baseline frequency of combined inappropriate behaviors (CI's) at 8 weeks, or when treatment goals are met | Baseline, up to eight weeks after first treatment visit
  Participants will be observed for CI's to evaluate the effectiveness of Desensitization

SECONDARY OUTCOMES:
Pediatric Eating Assessment Tool (PediEAT) | Baseline (pre-treatment), up to eight weeks (post-treatment)
  This is a parent-report instrument that is comprised of 78 questions that assess feeding difficulties across 4 subscales including: physiologic symptoms, problematic mealtime behaviors, selective/restrictive eating, and oral processing. Caregivers are asked to "think about what is typical for your child at this time" and to select from a scale of 6 response options including (0) Never, (1) Almost Never, (2) Sometimes, (3) Often, (4) Almost Always, and (5) Always. Higher scores indicate more symptoms of problematic feeding.
Family Management Measure of Feeding Questionnaire (FaMM Feed) | Baseline (pre-treatment), up to eight weeks (post-treatment)
  This is a 49 question survey that the parent/caregiver completes to evaluate mealtime feeding behaviors. Responses include: strongly disagree, disagree, neutral, agree, and strongly agree with each response score given is from 1-5 (1 = strongly disagree to strongly agree = 5). Lower scores indicating lower family management, or less feelings of being able to manage in the context of daily family life.
Parenting Stress Index-Short Form, 4th Edition (PSI4-SF) | Baseline (pre-treatment), up to eight weeks (post-treatment)
  This is a 36-item self-report questionnaire that assesses the level of stress in a parent-child relationship for parents of children 0-12 years of age. Each item is rated on a five-point Likert scale (1 = Strongly Agree, 2 = Agree, 3 = Not Sure, 4 = Disagree, and 5 = Strongly Disagree). It yields three subscales: Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC). Items are scored and added together to establish a total score as well as three subscale scores. The PSI-SF produces subscale raw scores ranging from 12 to 60 and an overall Parenting Stress (PSI-PS) total score that ranges from 36 to 180. Higher scores are indicative of a greater level of stress. A PSI-SF score above 85 indicates clinically significant parenting stress. The PSI-SF also includes a Defensive Responding (DR) scale to identify parents who might be attempting to minimize or deny problems.
Child Oral and Motor Proficiency Scale (ChOMPS) | Baseline (pre-treatment), up to eight weeks (post-treatment)
  This is a parent-report assessment of eating and drinking in children 6 months to 7 years. Consisting of 63-items, caregivers are asked to indicate the child's ability to perform a skill by choosing 'yes' (established skill; score = 2), 'sometimes' (emerging skill; score = 1), and 'not yet' (not yet emerging skill; score = 0). Total scores range from 0-126 with higher scores indicating greater skills. This measure yields 4 subscales including: basic movement patterns, fundamental oral-motor skills, oral-motor coordination, and complex movement patterns.
Child Behavior Checklist (CBCL) for ages 1 1/2 to 5 years old | Baseline (pre-treatment), up to eight weeks (post-treatment)
  The Checklist is a parent measure of emotional, behavioral and social problems in children ages 1.5-5 years. This 100-item measure yields broad-band scores of Internalizing Behavior Problems, Externalizing Behavior Problems, and Total Behavior Problems. It also yields eight additional problem scales: Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, and Aggressive Behavior. Caregivers rate each behavior or symptom on a three-point scale: not true (0), somewhat or sometimes true (1), or very true or often true (2). A computer program will be used to calculate the T-scores for each scale. Raw scores are converted to gender and age standardized scores (T-scores having a mean of 50 and SD of 10). Internal consistency Chronbach's alphas for each subscale are moderately high, ranging from .63 to .79. Alphas range from .78 to .97 for broad-band problem scales.
Child Behavior Checklist (CBCL) for ages 6-10 years old | Baseline (pre-treatment), up to eight weeks (post-treatment)
  The Checklist is a parent measure of emotional, behavioral and social problems in children ages 6-18 years. This 113-item measure yields broad-band scores of Internalizing Behavior Problems, Externalizing Behavior Problems, and Total Behavior Problems. It also yields eight additional problem scales: Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, and Aggressive Behavior. Caregivers rate each behavior or symptom on a three-point scale: not true (0), somewhat or sometimes true (1), or very true or often true (2). A computer program will be used to calculate the T-scores for each scale. Raw scores are converted to gender and age standardized scores (T-scores having a mean of 50 and SD of 10). Internal consistency Chronbach's alphas for each subscale are moderately high, ranging from .63 to .79. Alphas range from .78 to .97 for broad-band problem scales.
Change in Body Weight | Baseline (pre-treatment), up to eight weeks (post-treatment)
  Weight change from baseline
Change in Height | Baseline (pre-treatment), up to eight weeks (post-treatment)
  Height change from baseline
Change in Mid-upper arm circumference | Baseline (pre-treatment), up to eight weeks (post-treatment)
  Mid-upper arm circumference change from baseline
Change in Hand Grip Strength | Baseline (pre-treatment), up to eight weeks (post-treatment)
  Change in Hand Grip Strength from baseline will be measured using a JAMAR hydraulic hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Morris, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States